CLINICAL TRIAL: NCT00801099
Title: Benefit of a Single Preoperative Dose of Antibiotics in a Sub-Saharan District Hospital: Minimal Input, Massive Impact
Brief Title: Benefit of a Single Preoperative Dose of Antibiotics for the Prevention of Surgical Site Infections
Acronym: SSI2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Swiss Academy of Medical Sciences (SAMS) (Other)
Responsible Party: Prof. Dr. med. C. Hatz, Department of Medicine and Diagnostics, Swiss Tropical Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SSII
Record Dates: First submitted 2008-11-06; First posted 2008-12-03 (Estimated); Results first posted 2008-12-03 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-07

CONDITIONS: Surgical Site Infection
Keywords: Postoperative wound infection; surgical site infection; antimicrobial prophylaxis; developing countries; Sub-Saharan Africa; reduction of SSI using preoperative antibiotics
MeSH Terms: conditions — Surgical Wound Infection | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abx (Experimental): single shot dose of Amoxicillin/Clavulanic Acid approximately 30 min. preoperatively
  Interventions: Drug: Amoxicillin/Clavulanic Acid

INTERVENTIONS:
Drug: Amoxicillin/Clavulanic Acid — single shot dose of Amoxicillin/Clavulanic Acid approximately 30 min. preoperatively
  Other Names: Augmentin

SUMMARY:
In a rural hospital in Tanzania the rate of surgical site infections (SSI) was 21.6%. Inappropriate choice of antibiotics and of administration time were determined as sole risk factors in this setting. After implementation of a standardized procedure with a single shot dose of Amoxicillin/Clavulanic Acid approximately 30 min. preoperatively the rate of SSI dropped by 80% in spite of procedural risk factors like poor hygiene etc.

DETAILED DESCRIPTION:
Surgical Site Infections (SSIs) have an important socioeconomic impact prolonging the period of hospitalization and rehabilitation. Patients with SSIs are five times more likely to be readmitted and are even twice as likely to die compared to patients with similar interventions without SSI. In non-industrialized countries, the incidence of SSIs is higher and the consequences of SSI are even more severe: Many hospitals lack appropriate facilities for early diagnosis and treatment. In addition, microbiological identification of pathogens and susceptibility testing are rarely available, a prerequisite for targeted treatment of SSIs. Overcrowding and understaffing are additional risk factors for SSIs, common in these countries.

A study conducted at the local surgeons' suggestion in an 82-bed department of general surgery, obstetrics and gynecology, urology and orthopedics at the St. Francis Designated District Hospital (SFDDH) in Ifakara (Southern Tanzania) showed an SSI-rate of 21.6%.

The analyses of this study identified two major risk factors for SSI in clean and clean-contaminated surgical procedures: Inadequate timing of administration of routine antimicrobial prophylaxis (AMP) and inappropriate selection of antibiotics not covering the most commonly observed pathogens.

Therefore, an intervention study was discussed with the local surgeon in charge to improve selection and timing of routine AMP and thereby reduce the rate of SSIs.

The study design and objective were presented to all the staff during a general meeting and special duties and responsibilities discussed with the individual colleagues. Furthermore we distributed pocket flow sheets to the involved staff and hung up some laminated flow sheets in theatre.

ELIGIBILITY:
Inclusion Criteria:

* surgical patient
* clean or clean-contaminated surgery

Exclusion Criteria:

* infection
* preoperative antibiotic treatment
* postoperative antibiotic treatment
* open fractures

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2004-12; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christioph F Hatz, MD, Study Chair — Swiss Tropical & Public Health Institute
Locations (1):
- Swiss Tropical Institute, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Result] Saxer F, Widmer A, Fehr J, Soka I, Kibatala P, Urassa H, Frei R, Smith T, Hatz C. Benefit of a single preoperative dose of antibiotics in a sub-saharan district hospital: minimal input, massive impact. Ann Surg. 2009 Feb;249(2):322-6. doi: 10.1097/SLA.0b013e31819782fd. PMID 19212189

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All consecutive patients older than 15 years admitted for clean or clean-contaminated (according to Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for prevention of surgical site infection, 1999. Hospital Infection Control Practices Advisory Committee. Infect Control Hosp.Epidemiol. 1999;20:250-78) interventions.
Groups:
- Amoxicillin/Clavulanic Acid: Single shot dose of Amoxicillin/Clavulanic Acid approximately 30 minutes preoperatively.
Period: Overall Study
Arm/Group | Amoxicillin/Clavulanic Acid
Started | 276
Completed | 175
Not Completed | 101
Not completed — Lost to Follow-up | 101

BASELINE CHARACTERISTICS:
Arm/Group | Amoxicillin/Clavulanic Acid
Number analyzed (Participants) | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 230
  Male | 46
Region of Enrollment [Number; unit: participants]
  Tanzania | 276

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Surgical Site Infections
Time Frame: within 30 days postoperative
Measure: Number; unit: participants
Arm/Group | Amoxicillin/Clavulanic Acid
Number analyzed (Participants) | 175
participants | 11

2. Secondary Outcome: Sustainability of the Intervention in This Setting
Time Frame: during 3 month of study phase
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Amoxicillin/Clavulanic Acid
Serious Adverse Events (participants affected / at risk) | 11/276
Other Adverse Events (participants affected / at risk) | 0/276
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amoxicillin/Clavulanic Acid (N=276)
SSI (Surgical and medical procedures) | 11 — infection at surgical site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No